CLINICAL TRIAL: NCT04645836
Title: Impact of a Pharmacist-led Patient-centred Care Intervention Along With Text-Message Reminders, on the Management of Newly Diagnosed Tubercular Patients: a Protocol for a Randomized Controlled Trial'.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xi'an Jiaotong University (Other)
Collaborators: Pakistan Institute of Medical Sciences (Other Government); Quaid i Azam University Islamabad Pakistan (Unknown)
Responsible Party: Principal Investigator, Farman Ullah Khan, Principal Investigator (Phd Scholar), Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FUKhan
Record Dates: First submitted 2020-11-15; First posted 2020-11-27 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Pulmonary TB; TB
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Pharmaceutical Services

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): New management mode intervention: Pharmaceutical care A more recent strategy is pharmaceutical care, where a hospital provides timely patient education, monitoring and management of adverse drug reactions, identifying other drug-related problems, and an evaluation of treatment adherence by a clinical pharmacist. At the first visit, the clinical pharmacist provides a mobile phone number and encourages patients to contact them anytime if they need any consultation on the TB treatment.
  Short Message Service and Phone calls daily use of the mobile phone for a TB treatment will support pharmaceutical care. TB patients or family members will receive phone calls every evening (except Sunday) during the whole ambulatory TB treatment phase to assure that the patient takes the medication prescribed and provided by the TB physician and to collect information on treatment adherence and possible side effects.
  Interventions: Behavioral: New management mode
- No Intervention Group. (No Intervention): Treatment Group included in the control arm will receive traditional - clinical Directly Observed Therapy (DOT) as recommended by World Health Organization and routine treatment group (6 months treatment regimen); Routine health education provided by health care professionals.

INTERVENTIONS:
Behavioral: New management mode — New management mode intervention: Pharmaceutical care
  * SMS text messages and Phone Calls
  * Behavioural Educational leaflet
  * Self-Administered Therapy A financial incentive for mobile use
  Other Names: Pharmaceutical care, Mobile text, Financial incentive for mobile use
  Arms: Intervention Group

SUMMARY:
This project aims to standardize the management of "Pharmaceutical care with the two-way text messages and incentive for mobile usage during the treatment for tuberculosis patients, to improve the outcomes and compliance, reduce the risk of transmission and to evaluate the patient perspective in terms of their quality of life, shared decision making and satisfaction with services provided.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains a top ten leading cause of death globally despite it being a largely curable disease. New effective treatment supervision strategies are needed particularly in low-resource high TB burden settings and a potential solution is in the hands of nearly every patient - a mobile phone. Modern modular design mobile phone software applications ("apps") hold great promise to address this unmet need. Current technologies allow for rapid design modification based on end-user needs, implementation of native operating system (e.g., Android) versions for users with inconsistent internet access, and the integration of the patients' experiences with electronic health records using industry standards. Apps can perform multiple functions (e.g., automated reminders, symptom tracking, secure messaging, and multi-media education). Another strategy is pharmaceutical care which is utilized to enhance TB treatment compliance along with usage of mobile technologies, where clinical pharmacists provide patient education to improve the patient's knowledge on the disease and medication use and address the patient's drug-related problems. The use of a pharmaceutical care model to improve treatment outcomes and enhance adherence is on the rise in healthcare organizations. At the first visit, the clinical pharmacist provides a mobile phone number and encourages patients to contact them anytime if they need any consultation on the TB treatment. Patients will make prior arrangements with a study pharmacist to determine a convenient meeting place. These meetings will continue until treatment completion. To our knowledge, worldwide there has only been no randomized controlled trial (RCT) which has described the use of both pharmaceutical care model and two-way Short Message Service (SMS) communication with financial incentives (mobile money transfer cover healthcare costs related to SMS charges) to improve treatment outcomes. To find out both the pharmaceutical care model and two-way SMS communication with financial incentives would be helpful for TB patients in Pakistan. Therefore investigator aimed a study, to find out the effectiveness of trial gauged with the impact of the suggested model on the improved adherence, treatment completion, health-related quality of life and satisfaction with TB care.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Newly bacteriologically confirmed TB case (less than a month since diagnosis). This restriction (not more than one-month treatment) does not refer to patients whose most recent treatment outcome was a failure and who were assigned to a new treatment regimen.
* Own a mobile phone which operates on a telecom provider supported by our SMS platform
* Know how to and are able to receive SMS messages or Phone Call (Caretaker want to participate in case original patient do not participate)
* An address or residence location that is readily accessible for visiting, and willingness to inform the study team of any change of address during the treatment and follow-up period.
* No plans to move out of the catchment areas of the participating TB program sites within 9 months of enrollment.
* Facilities must have at least one TB doctor and one TB nurse available within the facility.
* Willingness to comply with study procedures and provide written informed consent prior to study enrollment.

Exclusion Criteria:

* Diagnosis is extra-pulmonary TB
* Currently enrolled in a clinical trial that prohibits enrollment in another study. Patients are leaving the area within the next six months.
* Patients are known at the start of treatment to require the treatment longer than it is recommended TB Management Guidelines for the appropriate type of TB.
* Previous history of TB, multidrug-resistant (MDR) or extensively drug-resistant (XDR) TB.
* Very ill patient's cognitive or physical disability that prevents full participation in the study such as vision, hearing, physically challenged, inability to swallow medications and unconscious Unable to answer questions.
* Pregnant females (treatment of TB infection will be deferred)
* Patients who are receiving treatment from private clinics (Who are not registered in the government TB sectors and they seek are form private health care facilities.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
TB treatment success rates | 6-9 Months
  TB treatment success rates defined by the World Health Organization. The investigators will compare clinically reported treatment outcomes between the intervention and control groups.
Adherence to treatment among drug-sensitive tuberculosis patients self reported and clinical record will checked for the follow up visits and drug taken | 6-9 Months
  Adherence Assessed daily from date of randomization until the date of a documented treatment outcome, up to 24 months after study enrollment date.Counting the number of administered pills, adequate adherence is more than 80% of administered pills.The measure adherence in TB patients for these determinations, we will measure patients' adherence via combined adherence endpoint consisting of Morisky Medication Adherence Scale and pill count rate.

SECONDARY OUTCOMES:
Health related Quality of Life of TB patients | 6-9 Months
  At baseline and upon completion of the treatment. To measure HRQoL (Health related Quality of Life) Revalidated data assortment tool European Quality of Life Scale EQ 5D 3L
Lost To Follow | 6-9 Months
  Lost to follow up or Treatment defaulters patients will be recorded from TB registers upon completion of the treatment
Patient satisfaction questionnaire | 6-9 Months
  At baseline and upon completion of the treatment. Satisfaction with information can be assessed with the satisfaction with information about medicines scale along with the Beliefs about medicines questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Fang, Phd, Study Chair — Xi'an Jiaotong University; Amjad Khan, Phd, Study Director — Quaid i Azam University Islamabad
Locations (1):
- Pakistan Institute of Medical Sciences Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Khan FU, Khan FU, Hayat K, Fang Y. Impact of a pharmacist-led patient-centred care intervention along with textmessage reminders, on the management of newly diagnosed tubercular patients: A protocol for a randomized controlled trial. Pak J Med Sci. 2024 Jan-Feb;40(3Part-II):487-491. doi: 10.12669/pjms.40.3.5356. PMID 38356837